CLINICAL TRIAL: NCT01960465
Title: Targeted Treatment of Obstructive Sleep Apnea to Reduce Cardiovascular Disparity
Brief Title: Race And CPAP Effectiveness
Acronym: RACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CLIN-022-13S
Record Dates: First submitted 2013-09-09; First posted 2013-10-10 (Estimated); Results first posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Sleep Apnea Syndromes
Keywords: CPAP treatment; hypertension
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypertension | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- African Americans (Experimental): 138 Self identified African American
  Interventions: Device: Continuous positive airway pressure
- non African Americans (Active Comparator): 53 Caucasians and 29 Other race (non African-Americans) Veterans.
  Interventions: Device: Continuous positive airway pressure

INTERVENTIONS:
Device: Continuous positive airway pressure — A portable ventilatory assist device, which is the standard first line treatment of sleep apnea.
  Other Names: CPAP

SUMMARY:
Obstructive sleep apnea (OSA) is a major public health problem in the U.S. and more than 35% of Veterans are at high risk for OSA. OSA is associated with progression of hypertension, an important health problem in Veterans. African Americans with OSA are at increased risk for poorly controlled hypertension and its health consequences. Implementing a care plan to increase the percentage of Veterans in whom blood pressure goals are achieved has been prioritized by Veterans Administration hospitals. Recent studies show that hypertension control can be improved with continuous positive airway pressure (CPAP) treatment of OSA. The aim of this proposal is to examine and compare the effects of CPAP treatment on 24-hour arterial blood pressure and central aortic blood pressure (measured non-invasively with a cuff on the upper arm) in African American and other Veterans.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) and hypertension are both common and severe problems in African American individuals (as noted in the International Society on Hypertension in Blacks consensus statement). CPAP treatment of OSA is effective in controlling hypertension in patients with OSA, but has not been studied in African Americans, a high-risk population with potentially large health gains. This is an area of significance because poorly controlled hypertension leads to progression of cardiovascular disease (CVD) and morbidity in this population. By identifying CPAP treatment-response and relevant moderators of this response in African Americans with hypertension and OSA, targeted treatment of OSA can be implemented, reducing the excess burden of CVD. The investigators will determine the relative magnitude of hypertension response to CPAP treatment (ambulatory blood pressure and central aortic blood pressure) in 220 African American and Veterans of other race(s) with hypertension and newly diagnosed OSA (specific aim 1). The investigators will measure changes in pathogenic biomarkers (urinary cumulative sympathetic nervous system activity and oxidative stress) that are responsive to CPAP treatment in addition to hypertension assessments. Further, the investigators will examine the role of excessive daytime sleepiness (EDS), a potentially important moderator of treatment response, in these two patient populations (specific aim 2). Finally, the investigators will adjust the outcomes assessment for the anticipated biological heterogeneity among self-identified African Americans by measuring genetic ancestry (exploratory aim). This award will provide the foundation for the goals of this research program to reduce CVD disparity in diverse populations with targeted treatment of OSA.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified African American and other Veterans (of self-identified race other than African American)
* Age: 30-70 years
* Hypertension
* Apnea hypopnea index (AHI) 15/hour on home sleep apnea test

Exclusion Criteria:

* Past/current treatment of Obstructive Sleep Apnea or other primary sleep disorders
* Active uncontrolled medical conditions
* Shift work in past 6 months
* Current drug use
* Pregnancy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bharati Prasad, MD, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (1):
- Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Imayama I, Gallagher C, Grand J, Follman B, Kansal M, Prasad B. Defining the impact of continuous positive airway pressure therapy on diastolic function in adults with moderate-to-severe obstructive sleep apnea. J Sleep Res. 2023 Aug;32(4):e13856. doi: 10.1111/jsr.13856. Epub 2023 Feb 26. PMID 36843239
- [Derived] Imayama I, Gupta A, Yen PS, Chen YF, Keenan B, Townsend RR, Chirinos JA, Weaver FM, Carley DW, Kuna ST, Prasad B. Socioeconomic status impacts blood pressure response to positive airway pressure treatment. J Clin Sleep Med. 2022 May 1;18(5):1287-1295. doi: 10.5664/jcsm.9844. PMID 34931603

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2015 to August 2019, recruitment by chart review (results of home sleep apnea test) at Jesse Brown VA.
  Participants were contacted by phone, consented on screening/Visit 1.
Pre-assignment Details: All participants had moderate to severe newly diagnosed/untreated OSA> They were started on PAP therapy after visit 1.
Period: Overall Study
Arm/Group | African Americans | Non African Americans
Started | 138 | 82
Completed | 118 | 73
Not Completed | 20 | 9

BASELINE CHARACTERISTICS:
Population: Analysis population consisted of 191 participants, after accounting for drop-out and missing data for primary outcome of 24-hour BP.
Groups:
- Total: Total of all reporting groups
Arm/Group | African Americans | Non African Americans | Total
Number analyzed (Participants) | 138 | 82 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.74 (10.3) | 53.1 (10.4) | 53.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 26
  Male | 121 | 73 | 194
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 138 | 0 | 138
  White | 0 | 53 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 29 | 29
Region of Enrollment [Number; unit: participants]
  United States | 138 | 82 | 220
24 hour blood pressure [Mean (Standard Deviation); unit: mm Hg] | 130.55 (13.9) | 126.49 (13.6) | 129.02 (13.9)

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Ambulatory Blood Pressure
Description: Mean systolic and diastolic blood pressure measured over 24 hours with ambulatory monitor (Spacelabs).
  The change in blood pressure values were calculated as 3 months BP - baseline BP.
  The mean and standard deviation in the sample are noted below.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Non African Americans: 82 Other race (non African Americans) Veterans.
  Continuous positive airway pressure: A portable ventilatory assist device, which is the standard first line treatment of sleep apnea.
Arm/Group | African Americans | Non African Americans
Number analyzed (Participants) | 118 | 73
mm Hg
  Systolic BP | -1.93 (13) | -0.64 (7.6)
  Diastolic BP | -1.38 (9.3) | -1.19 (7.9)

2. Secondary Outcome: Central Aortic Blood Pressure
Description: Central aortic blood pressure (CABP) measured noninvasively with a cuff (SphygmoCor XCEL).
  The change in CABP values were calculated as 3 months CABP - baseline CABP. The mean and standard deviation in the sample are noted below.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: m/sec and percent
Arm/Group | African Americans | Non African Americans
Number analyzed (Participants) | 118 | 73
m/sec and percent
  Pulse Wave Velocity | -0.20 (2.0) | -0.23 (1.6)
  Augmentation Index | -1.20 (10.6) | -0.68 (10.7)

3. Secondary Outcome: Urinary Sympathetic Activity (Catecholamines) and Oxidative Stress (8-isoprostane)
Description: Urine samples from participants over 24 hours will be analyzed for catecholamines and overnight sample will be partitioned for measurement of oxidative stress.
  The change in urine catecholamine values were calculated as 3 months - baseline.
  The mean and standard deviation in the sample are noted below.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ng/mg creatinine
Arm/Group | African Americans | Non African Americans
Number analyzed (Participants) | 118 | 73
ng/mg creatinine
  Urine Epinephrine | 0.02 (1.8) | -0.26 (1.4)
  Urine Norepinephrine | -3.7 (12.2) | -2.7 (11.1)

ADVERSE EVENTS:
Time Frame: 3-5months.
Description: AE and SAE definitions used were consistent with clinicaltrials.gov.
Arm/Group | African Americans | Non African Americans
All-Cause Mortality (participants affected / at risk) | 0/138 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/138 | 0/82
Other Adverse Events (participants affected / at risk) | 0/138 | 0/82

LIMITATIONS AND CAVEATS:
The limitations of the study are as follows: Lower than anticipated enrollment of Whites & lower than anticipated adherence to CPAP therapy overall, particularly in African American Veterans.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT01960465/Prot_SAP_000.pdf